CLINICAL TRIAL: NCT02127957
Title: Effects of a Program of Aerobic and Resistance Exercises Combined in Patients With Cystic Fibrosis (CF) With Impaired Glucose Tolerance or Diabetes Related to CF Without Medication
Brief Title: Effects of an Exercise Program Among CF Patients With Dysglycemia
Acronym: FKEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Yves Berthiaume, Dr Yves Berthiaume,, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: FKEX_12.356
Record Dates: First submitted 2014-04-18; First posted 2014-05-01 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis Related Diabetes
Keywords: cystic fibrosis; exercise; Cystic fibrosis related diabetes
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Other): Exercise group will have 6 visit and 8 phone call. Subject will have to do prescribed exercice for 1h, 3 times a week for 12 weeks.
  Interventions: Other: Exercise
- Control (No Intervention): Control group will have 4 visit and 3 phone call. They will receive standard counselling for exercise in cystic fibrosis, but no prescribed exercice will be given.

INTERVENTIONS:
Other: Exercise — Exercise will be prescribed by kinesiologist and will be done 3 times a week for 1 hour by subject. Every 4 weeks subject will be on supervised training session.
  Arms: Exercise

SUMMARY:
The objective of the investigators research program is to determine whether a combined exercise program (aerobic and resistance) improves abnormal glucose tolerance and diabetes control in CF patients. This program of exercises to increase strength and muscle endurance, exercise tolerance, will be assessed in a group of 12 CF patients with impaired glucose tolerance. The effect of exercise will be compared with a control group of 12 patients also glucose intolerant but do not participate in structured physical activity program. The duration of the exercise program will be 12 weeks and several measures (glucose tolerance, inflammatory profile, lung function, exercise capacity, muscle strength and endurance) will be conducted pre and post program to assess the program's impact .

DETAILED DESCRIPTION:
A total of 24 subjects with CF with impaired glucose tolerance or with diabetes related to CF (CFRD) unmedicated will be recruited. Participants will be recruited through a research nurse in CF , which will analyze the available data to medical records and seek the participation of subjects who meet the inclusion and exclusion criteria . Patients receive during their visit to the outpatient clinic of FK at Hotel -Dieu du CHUM hospital , a inform consent form (ICF) for the study. Their intention to participate and the main inclusion and exclusion criteria will be confirmed in a telephone interview conducted by a member of the team at the IRCM. Finally, during the visit at the IRCM , the subject will get answer to his question for ICF and ICF will be signed before any procedure.

All participants who agree to participate in the research project must undergo a short telephone interview (20 minutes) and 4 assessment visits ( approximately 1-5 hours) Pre (2 visits ) and post (2 visits ) study . The control patients with delayed exercises conduct a further assessment visit at the end of the training.

GROUP 1 EXERCISES : Patients in exercises group will be required to take part of two supervised training sessions and 8 follow up phone call . The exercise program will be performed three times per week for about one hour .

GROUP 2 CONTROL: Participants in the control group will be contacted by phone once a month following entry into the study. On this occasion a reminder to complete the physical activity log will be realized. Following the visit #6 , patients in the control group will be invited to participate in a second study phase to participate in supervised exercise program . This participation will involve an additional 12 weeks of follow-up, which included the same visit as Group 1 with exercises. In this case, to simplify participation and reduce the volume of blood collected , the final visit (#5) of the project will also be the first visit of exercises phase. This part of study, involves 2 supervised training sessions and 8 follow up phone call . The exercises program will be performed three times per week for about one hour .

ELIGIBILITY:
Inclusion Criteria :

* Men or women 18 years and older.
* Diagnosis of CF documented.
* Obstructive ventilatory deficit light to moderate , as defined in the guidelines of the ATS / ERS , an FEV / FVC ratio > 70% and ≥ 40% FEV .
* Stable health status, no episode of superinfection in the past 6 weeks.
* Impaired glucose tolerance , glucose > 11.1 mmol / L at the 1st hour of the OGTT or unmedicated CFRD.
* Patients who wants to participate in an exercise program for 12 weeks.
* Sedentary (less than 105 min / week of physical activity ) .

Exclusion Criteria :

* Exacerbation of respiratory symptoms with or without hospitalization , or use of oral antibiotics in the last 6 weeks.
* Exacerbation with intravenous antibiotics .
* Severe obstructive deficit as defined by FEV <40% , with an FEV / FVC ratio <70 %.
* Any other disease or condition that may limit exercise performance .
* Without treatment with oral hypoglycemia , insulin, oral anti -inflammatory and other treatments that may influence glucose metabolism (patient under cortef accepted) .
* Hemoptysis ( > 50-60 cc) in the last 6 weeks.
* Desaturation during exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in glycemia at 2h of -1.5 mmol/L | baseline and week 13
  Evaluate if patient with CF have improved glucose tolerance at the second hour of a Oral glucose tolerance test (OGTT) following a combined exercise program.

SECONDARY OUTCOMES:
inflammatory marker change | baseline and week 13
  Assess whether the practice of regular combined physical activity program modifies the inflammatory profile (C-reactive protein, cytokines (IL-1β, IL-13, IL-6, IL-8, IL-10, TNF, CH3Li)) associated with CF diabetes.
VO2max changes | baseline and week 13
  Evaluate if regular combined physical activity program improves exercise tolerance in CF patient.
muscular strength | baseline and week 13
  Evaluate if regular combined physical activity program improves muscle strength and endurance.
area under the insulin curve | basline and week 13
  Evaluate if regular combined physical activity program improves insulin sensitivity.
Changes in glycemia of -1.5mmol/L at 1h | basline and week 13
  Evaluate if regular combined physical activity program improves glucose tolerance at one hour of the OGTT.
quality of life changes | baseline and week 13
  Evaluate if regular combined physical activity program improves quality of life in CF.
lean mass changes | basline and week 13
  Evaluate if regular combined physical activity program improves lean mass in CF.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Berthiaume, Md, Principal Investigator — Institut de Recherches Cliniques de Montreal; Remi Rabasa-Lhoret, Md, Study Chair — Institut de Recherches Cliniques de Montreal
Locations (1):
- CRIMontreal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Beaudoin N, Bouvet GF, Coriati A, Rabasa-Lhoret R, Berthiaume Y. Combined Exercise Training Improves Glycemic Control in Adult with Cystic Fibrosis. Med Sci Sports Exerc. 2017 Feb;49(2):231-237. doi: 10.1249/MSS.0000000000001104. PMID 27669451